CLINICAL TRIAL: NCT04819620
Title: A Randomised, Double-Blind, Placebo-controlled Study of Single and Multiple Ascending Doses of PN-232 in Healthy Volunteers
Brief Title: Pharmacokinetics of PN-232 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: PN-232-01
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Single Dose (Experimental): Single dose administration
  Interventions: Drug: PN-232; Drug: Placebo
- Multiple Dose (Experimental): Multiple dose administration
  Interventions: Drug: PN-232; Drug: Placebo
- Solid Dose Comparison (Experimental): Solid dose administration
  Interventions: Drug: PN-232

INTERVENTIONS:
Drug: PN-232 — Active Drug
Drug: Placebo — Matching Placebo
  Arms: Multiple Dose; Single Dose

SUMMARY:
This Phase 1 study is designed to determine the safety, tolerability and pharmacokinetics of PN-232 in healthy volunteers. It is a first-in-human (FIH) study for PN-232 that will be conducted in three parts. Part 1 is a single ascending dose study, Part 2 is multiple ascending dose study, and Part 3 is crossover solid dose comparison and effect of food study.

DETAILED DESCRIPTION:
Part 1: Approximately 32 subjects will be enrolled into 4 cohorts to receive PN-232 or placebo as single doses.

Part 2: Up to 40 subjects will be enrolled into 4 cohorts to receive PN-232 or placebo once daily for 10 days.

Part 3: Twelve subjects will receive single doses of PN-232 in a 3-way, randomized, crossover fashion.

In total, approximately 84 subjects will participate.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects must have BMI between 18 and 32 kg/m2
* Subjects must be non-smokers or social smokers
* Subjects must comply with contraception requirements
* Subjects must be willing to consume meals provided by the clinical center
* Subjects must be willing to attend required clinic visits
* Subjects must be suitable candidates for study procedures

Key Exclusion Criteria:

* Subject with a history of clinically significant endocrine, neurological, cardiovascular, hematological, hepatic, immunological, renal, respiratory, gastrointestinal or genitourinary abnormalities or diseases within previous 10 years
* Subjects with a history of surgical resection of the stomach, small or large intestine
* Subjects with a fever or symptomatic viral or bacterial infection within 2 weeks of screening or intestinal infection within 30 days prior to screening
* Subjects with clinically significant laboratory abnormalities
* Subjects with corrected QT greater than 450 msec in males and 470 msec in females
* Subjects who test positive for Hepatitis C or B, or HIV at Screening
* Subjects who cannot refrain from use of prescription and non-prescription drugs and herbal remedies prior to initial dose of study drug and throughout the study
* Subjects who test positive for drugs of abuse or alcohol at Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Safety of PN-232 | 10 days
  Number and Severity of Adverse Events

SECONDARY OUTCOMES:
Peak concentration of PN-232 in plasma | 10 days
  Peak concentration (Cmax) of PN-232
Area under the Concentration (AUC) of PN-232 | 10 days
  AUC over 24 hours on Day 10 for PN-232

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Protagonist Clinical Site, Adelaide, South Australia
  - Protagonist Study Site, Nedlands, Western Australia